CLINICAL TRIAL: NCT03664544
Title: An Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of MCI-186 in Subjects With Severe Hepatic Impairment Compared to Subjects With Normal Hepatic Function
Brief Title: PK Study in Subjects With Severe Hepatic Impairment
Acronym: MCI-186-E05 HP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MCI-186-E05; 2018-001163-23 (EudraCT Number)
Record Dates: First submitted 2018-08-27; First posted 2018-09-10 (Actual); Results first posted 2020-04-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Severe Hepatic Impairment; Healthy
Keywords: Severe Hepatic Impairment; Healthy
MeSH Terms: interventions — Edaravone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subjects with severe hepatic impairment (Experimental): HP PK MCI-186
  Interventions: Drug: MCI-186
- Subjects with normal hepatic function (Experimental): NHV PK MCI-186
  Interventions: Drug: MCI-186

INTERVENTIONS:
Drug: MCI-186 — 30 mg MCI-186 will be administered intravenously over 60 minutes.
  Other Names: Edaravone; Radicava; Radicut

SUMMARY:
This is an open-label, single-dose study in male and female subjects with severe hepatic impairment and in male and female subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

All subjects

* 1. Able to provide written informed consent to participate in this study after reading the participant information sheet and Informed Consent Form (ICF), and after having the opportunity to discuss the study with the Investigator or designee.
* 2. Male or female subjects age 18 to 75 years (inclusive) at signature of the ICF.
* 3. In the Investigator's opinion, subject is able to understand the nature of the study and any risks involved in participation, and willing to cooperate and comply with the Protocol restrictions and requirements.
* 4. A body weight of ≥50 kg and a body mass index (Quetelet index) ranging from 18 to 37 kg/m2 (inclusive) at Screening and Day -1.
* 5. Female subjects who are:

  1. postmenopausal for at least 1 year, confirmed by follicle-stimulating hormone assessment (>40 mIU/mL), or
  2. surgically sterilised (hysterectomy, bilateral oophorectomy or salpingectomy), or
  3. congenital sterility. Female subjects of child-bearing potential must practice effective contraception (see Protocol body) from the Screening Visit or at least 2 weeks before IMP administration, until 30 days after IMP dosing. Male subject must practice effective contraception from the time of IMP dosing until 90 days after IMP dosing. Adhering to strict abstinence is considered an accepted contraceptive method.

Hepatic impaired subjects (in addition)

* 6. Diagnosis of cirrhosis due to parenchymal liver disease, which is documented in the medical history and physical examination and confirmed by at least one of the following: hepatic ultrasound, computed axial tomography scan, magnetic resonance imaging and/or liver biopsy. A Child-Pugh classification score of 10 to 14 obtained during the Screening period (i.e., within 21 days of IMP administration).
* 7. Chronic (>6 months) and stable hepatic impairment defined as no clinically significant change in disease status at least 14 days before Screening.
* 8. Acceptable clinical conditions in the opinion of the Investigator on the basis of a physical examination, medical history, 12-lead electrocardiogram (ECG), vital signs and clinical laboratory tests (biochemistry, haematology, coagulation and urinalysis) at Screening, Day -1 and pre-dose on Day 1. Subjects with stable mild chronic concurrent diseases, such as degenerative joint disease, controlled diabetes, hypertension or hyperlipidaemia, etc. may be included.

Healthy subjects (in addition)

* 9. Subjects with normal hepatic function confirmed with tests within the normal reference range or results with minor deviations which are not considered by the Investigator to be clinically significant.
* 10. Good health and free from clinically significant illness or disease in the opinion of the Investigator on the basis of a physical examination, medical history, ECG, vital signs and clinical laboratory tests (biochemistry, haematology, coagulation and urinalysis) at Screening, Day -1 and pre-dose on Day 1.

Exclusion Criteria:

All subjects

* 1. Presence or history of severe allergy to food, or any medical product or relevant excipient that is of clinical significance.
* 2. Subjects who have previously been administered MCI-186.
* 3. As a result of the medical screening process, the Investigator considers the subject not suitable for the study.
* 4. Clinically significant 12-lead ECG abnormalities, including but not limited to, corrected QT interval using Fridericia's formula (QTcF) of >450 ms (male subjects) or >470 ms (female subjects) at Screening, Day -1 or before dosing.
* 5. Any other history or condition (surgical or medical) of disease which will increase the risk to the subject, will affect the PK of the study drug, or will otherwise influence the assessments to be made in this study, in the opinion of the Investigator. Subjects who have undergone cholecystectomy may be included.
* 6. History of drug abuse or tested positive for alcohol or drugs of abuse at Screening and Day -1, excluding drugs which may cause a positive drug or abuse test if medically indicated or prescribed.
* 7. Subjects who regularly, or on average, drink more than 35 units of alcohol per week (one unit is equivalent to 300 mL of beer, 25 mL of spirits or 150 mL of wine).
* 8. Presence of active infection requiring antibiotics.
* 9. Positive test for human immunodeficiency virus antigen/antibody at Screening.
* 10. Donation of one or more units of blood (450 mL) within 3 months prior to Screening, or plasma in the 7 days prior to Screening, or platelets in the 6 weeks prior to Screening, or the intention to donate blood within 3 months after the last Follow-up assessment.
* 11. Participation in another study within the last month (if single dose), or at least 4 months (if multiple dose), or within 10 times the half-life of the respective drug (whichever is longer) before Screening. For biologics, the minimum period is at least 6 months before Screening, the period of the pharmacodynamic effect, or 10 times the half life of the respective drug, whichever is longer.
* 12. Subject is currently taking non-permitted concomitant medication. The subjects with normal hepatic function are restricted from use of any concomitant medications (including paracetamol) unless discussed and agreed with the Sponsor. In subjects with hepatic impairment, the use of prescribed medications is permitted for hepatic or concomitant disease as described in the Protocol body.
* 13. Not willing to abstain from consumption of coffee, tea, cola, energy drinks or chocolates from admission to the unit (Day -1) to discharge from the unit (Day 3).
* 14. Uncontrolled, or untreated hypertension defined as a mean of three repeated measurements of systolic blood pressure >180 mmHg and/or diastolic blood pressure >100 mmHg.
* 15. Subjects have estimated glomerular filtration rate <60 mL/min/1.73 m2 as determined by Modification of Diet in Renal Disease formula.
* 16. Any condition associated with dehydration.
* 17. Female subjects:

  1. who have a positive pregnancy test at Screening or on Day -1.
  2. who are pregnant, lactating or planning to become pregnant during the study.

Hepatic impaired subjects (in addition)

* 18. Subjects with severe ascites or pleural effusion which will, in the opinion of the Investigator, adversely affect the subject's ability to participate in the study.
* 19. Subjects with severe encephalopathy (Grade III or IV).
* 20. Subjects with sclerosing cholangitis.
* 21. Serum albumin <2.0 g/dL.
* 22. Haemoglobin <10 g/dL.
* 23. Start of any new medication or any changes to a current dosage within 14 days before IMP administration.

Healthy subjects (in addition)

* 24. History or presence of any parenchymal hepatic disease.
* 25. Positive test for hepatitis B surface antigen or hepatitis C virus antibody.
* 26. History of or active suicidal ideation, or suicide attempt as evidenced by positive response to either Question 4 (active suicidal ideation with some intent to act) or Question 5 (active suicidal ideation with specific plan and intent) on the Columbia-Suicide Severity Rating Scale (C-SSRS; Screening Version).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Mitsubishi Tanabe Pharma Europe Ltd
Locations (3):
- Investigational Centre, Prague, Czechia
- Investigational Centre, Miskolc, Hungary
- Investigational Centre, Bratislava, Slovakia

REFERENCES:
- [Derived] Nakamaru Y, Kakubari M, Yoshida K, Akimoto M, Todorovic V, Greis T, Kondo K. Open-label, Single-dose Studies of the Pharmacokinetics of Edaravone in Subjects with Mild, Moderate, or Severe Hepatic Impairment Compared to Subjects with Normal Hepatic Functioning. Clin Ther. 2020 Aug;42(8):1467-1482.e4. doi: 10.1016/j.clinthera.2020.06.016. Epub 2020 Aug 14. PMID 32800532

RESULTS

PARTICIPANT FLOW:
Groups:
- HP PK MCI-186: Subjects with severe hepatic impairment (A Child-Pugh classification score of 10 to 14) were intravenously administered 30 mg MCI-186 over 60 minutes on the morning of Day 1.
- NHV PK MCI-186: Subjects with normal hepatic function were intravenously administered 30 mg MCI-186 over 60 minutes on the morning of Day 1
Period: Overall Study
Arm/Group | HP PK MCI-186 | NHV PK MCI-186
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | HP PK MCI-186 | NHV PK MCI-186 | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (7.9) | 53.0 (8.0) | 57.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameters of MCI-186: Peak Drug Concentration (Cmax)
Description: Unchanged MCI-186
Time Frame: Day 1 to 3 (Pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h)
Population: PK population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | HP PK MCI-186 | NHV PK MCI-186
Number analyzed (Participants) | 6 | 6
ng/mL | 347.6 (146.8) | 280.3 (101.0)

2. Primary Outcome: Pharmacokinetic Parameters of MCI-186: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-last)
Description: Unchanged MCI-186
Time Frame: Day 1 to 3 (Pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h)
Population: PK population
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | HP PK MCI-186 | NHV PK MCI-186
Number analyzed (Participants) | 6 | 6
h*ng/mL | 473.90 (163.28) | 394.65 (160.01)

3. Primary Outcome: Pharmacokinetic Parameters of MCI-186: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-∞)
Description: Unchanged MCI-186
Time Frame: Day 1 to 3 (Pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h)
Population: PK population
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | HP PK MCI-186 | NHV PK MCI-186
Number analyzed (Participants) | 6 | 6
h*ng/mL | 496.98 (183.81) | 416.34 (164.96)

4. Secondary Outcome: Incidence of Adverse Events (AEs) and Serious Adverse Events
Description: Number of adverse events
Time Frame: Day -1 to Day 7
Population: Safety Analysis Set
Measure: Number; unit: Events
Arm/Group | HP PK MCI-186 | NHV PK MCI-186
Number analyzed (Participants) | 6 | 6
Events
  Adverse events | 0 | 1
  Serious adverse events | 0 | 0
  Treatment emergent adverse events | 0 | 1
  Adverse Drug reaction | 0 | 1
  TEAE leading to discontinuation of study drug | 0 | 0

5. Secondary Outcome: Pharmacokinetic Parameters of MCI-186: Half-life (t½)
Description: Unchanged MCI-186
Time Frame: Day 1 to 3 (Pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h)
Population: PK population
Measure: Mean (Standard Deviation); unit: h
Arm/Group | HP PK MCI-186 | NHV PK MCI-186
Number analyzed (Participants) | 6 | 6
h | 3.88 (1.12) | 9.51 (6.62)

6. Secondary Outcome: Pharmacokinetic Parameters of MCI-186: Time to Reach Peak Concentration (Tmax)
Description: Unchanged MCI-186
Time Frame: Day 1 to 3 (Pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h)
Population: PK population
Measure: Median (Full Range); unit: h
Arm/Group | HP PK MCI-186 | NHV PK MCI-186
Number analyzed (Participants) | 6 | 6
h | 1.02 [0.25 to 1.05] | 1.02 [1.00 to 1.03]

7. Secondary Outcome: Pharmacokinetic Parameters of MCI-186: Terminal Elimination Rate Constant (λZ)
Description: Unchanged MCI-186
Time Frame: Day 1 to 3 (Pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h)
Population: PK population
Measure: Mean (Standard Deviation); unit: /h
Arm/Group | HP PK MCI-186 | NHV PK MCI-186
Number analyzed (Participants) | 6 | 6
/h | 0.19 (0.06) | 0.15 (0.14)

8. Secondary Outcome: Pharmacokinetic Parameters of MCI-186: Total Clearance (CL)
Description: Unchanged MCI-186
Time Frame: Day 1 to 3 (Pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h)
Population: PK population
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | HP PK MCI-186 | NHV PK MCI-186
Number analyzed (Participants) | 6 | 6
L/h | 66.82 (21.49) | 78.72 (20.51)

9. Secondary Outcome: Pharmacokinetic Parameters of MCI-186: Volume of Distribution at Steady State (Vss)
Description: Unchanged MCI-186
Time Frame: Day 1 to 3 (Pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h)
Population: PK population
Measure: Mean (Standard Deviation); unit: L
Arm/Group | HP PK MCI-186 | NHV PK MCI-186
Number analyzed (Participants) | 6 | 6
L | 133.86 (71.05) | 449.79 (438.26)

10. Secondary Outcome: Pharmacokinetic Parameters of MCI-186: Volume of Distribution During the Terminal Phase (VZ)
Description: Unchanged MCI-186
Time Frame: Day 1 to 3 (Pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h)
Population: PK population
Measure: Mean (Standard Deviation); unit: L
Arm/Group | HP PK MCI-186 | NHV PK MCI-186
Number analyzed (Participants) | 6 | 6
L | 359.85 (130.06) | 1064.88 (888.10)

11. Secondary Outcome: Pharmacokinetic Parameters of MCI-186: Mean Residence Time (MRT)
Description: Unchanged MCI-186
Time Frame: Day 1 to 3 (Pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h)
Population: PK population
Measure: Mean (Standard Deviation); unit: h
Arm/Group | HP PK MCI-186 | NHV PK MCI-186
Number analyzed (Participants) | 6 | 6
h | 2.27 (1.87) | 5.51 (4.60)

12. Secondary Outcome: Pharmacokinetic Parameters of MCI-186: Unbound Area Under the Concentration-time Curve From Time Zero to Infinity (AUCu0-∞)
Description: Unchanged MCI-186
Time Frame: Day 1 to 3 (Pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h)
Population: PK population
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | HP PK MCI-186 | NHV PK MCI-186
Number analyzed (Participants) | 6 | 6
h*ng/mL | 65.41 (28.71) | 45.33 (13.97)

13. Secondary Outcome: Pharmacokinetic Parameters of MCI-186: Unbound Total Clearance (Clu)
Description: Unchanged MCI-186
Time Frame: Day 1 to 3 (Pre-dose, 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h and 48h)
Population: PK population
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | HP PK MCI-186 | NHV PK MCI-186
Number analyzed (Participants) | 6 | 6
L/h | 529.83 (200.93) | 702.10 (159.63)

ADVERSE EVENTS:
Time Frame: Day -1 to Day 7
Arm/Group | HP PK MCI-186 | NHV PK MCI-186
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HP PK MCI-186 (N=6) | NHV PK MCI-186 (N=6)
Sinus Bradycardia (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT03664544/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT03664544/SAP_001.pdf